CLINICAL TRIAL: NCT04770987
Title: Lateral Neck Flexor Endurance in Individuals With and Without Systemic Hyperlaxity
Brief Title: Lateral Neck Flexor Endurance and Hyperlaxity
Status: Completed | Type: Observational
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Other Study IDs: PRO02021000205
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Physical Endurance; Hypermobility, Joint; Muscular Weakness
Keywords: neck musculature; endurance; tests and measures
MeSH Terms: conditions — Joint Instability; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hyperlaxity: 30 individuals with systemic hyperlaxity as defined by a score of 5 or greater on the Beighton Hypermobility Scale
  Interventions: Other: lateral neck flexor endurance test
- control: 30 healthy, age and gender matched individuals without hyperlaxity
  Interventions: Other: lateral neck flexor endurance test

INTERVENTIONS:
Other: lateral neck flexor endurance test — Individuals will maintain the head in a neutral position off the ground in sidelying for as long as possible.

SUMMARY:
The lateral neck flexor endurance test has been proposed to assess for unilateral muscular deficits. It is not known if individuals with hyperlaxity have different muscular endurance than individuals without hyperlaxity.

DETAILED DESCRIPTION:
Thirty individuals with systemic hyperlaxity as determined with the Beighton scale will be assessed for lateral neck flexor endurance and compared to age and gender matched controls. Basic demographic information will be collected, and all individuals will report Neck Disability Index (NDI) and Numeric Pain Rating Scales (NPRS) for their neck, as well duration of any neck pain. All participants will then undergo testing of lateral neck flexor muscle endurance, repeated twice on each side. Average hold times will be compared for individuals with hyperlaxity (5 or greater on Beighton scale) and the healthy age and gender matched controls. Analysis will also include covariates of NDI scores, pain scores, and chronicity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

systemic hyperlaxity of 5 or greater on Beighton Index, healthy age/gender matched controls

Exclusion Criteria:

* neck pain that spreads into the arms;
* whiplash injury within the last 6 weeks;
* diagnosed neuropathy or other nervous system disorders;
* a history of spinal surgery in their neck;
* fibromyalgia;
* insulin dependent diabetes;
* involved in legal activity regarding neck pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals between the ages of 18-60 with and without systemic hyperlaxity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
lateral neck flexor endurance | single testing session at enrollment
  maximum hold time

SECONDARY OUTCOMES:
Beighton Hyperlaxity Scale | at enrollment
  Assessment of systemic hyperlaxity, 0-9 points, higher indicates greater hyperlaxity
Neck Disability Index | at enrollment
  Questionnaire assessing impact of neck symptoms on function, 0-100 points, higher score indicates greater disability
Numeric pain rating scale | at enrollment
  assessment of neck pain, 0-10 with higher indicating greater levels of pain

CONTACTS AND LOCATIONS:
Overall Officials: Brian Swanson, PT, DSc, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No